CLINICAL TRIAL: NCT03490435
Title: Diagnostics of Intestinal Parasitosis in Inhabitants of Kuyavian-Pomeranian Province in Poland
Brief Title: Intestinal Parasites in Inhabitants of Kuyavian-Pomeranian Province in Poland
Status: Completed | Type: Observational
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Paweł Sutkowy, Assistant professor, Nicolaus Copernicus University
Other Study IDs: KB 765/2016
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Intestinal Disease, Parasitic; Chronic Disease
Keywords: Per os invasions; Giardiasis; Toxoplasmosis; Taeniasis; Cryptosporidiosis; Trichinosis; Ascariasis; Echinococcosis
MeSH Terms: conditions — Intestinal Diseases, Parasitic; Chronic Disease; Giardiasis; Toxoplasmosis; Taeniasis; Cryptosporidiosis; Trichinellosis; Ascariasis; Echinococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: Both healthy and ailing individuals, both sex, including adults and children.
  Interventions: Diagnostic Test: Tests for diagnosis of intestinal parasitic diseases

INTERVENTIONS:
Diagnostic Test: Tests for diagnosis of intestinal parasitic diseases — Feces testing:
  1. fresh fecal samples will be used to preparing direct (saline and iodine wet) mounts using supplementary techniques (flotation, sedimentation), as well as temporary mounts (hematoxylin and trichrome staining). Other technique of fresh fecal samples examination will be ParaSys™
  2. A non-preserved stool samples will be stored below -20°C. Defrosted fecal specimen will be subjected to enzyme-linked immunosorbent assays (ELISA) - Giardia antigen test (coproantigens)

SUMMARY:
The goal of the proposed study is to assess the prevalence of intestinal parasitic diseases in adults and children. These invasions are included to "dirty hand diseases" (per os invasions), therefore it applies mainly preschool children.

DETAILED DESCRIPTION:
It is estimated that 75% of the world's population is infected with parasites and although parasitic diseases are mostly observed in the poor tropical and subtropical countries, there are also many diseases caused by parasites in Poland. In Poland, particular attention is paid to the following parasitic diseases closely related to the digestive system: giardiasis, taeniasis (including cysticercosis), ascariasis, cryptosporidiosis, toxoplasmosis, trichinosis, echinococcosis.

Symptoms of such invasions may include: allergic rhinitis of unknown origin, chronic fatigue or food intolerance. Moreover, many of them are asymptotic, therefore the study group will consist of both healthy people and individuals with undiagnosed diseases or/and chronic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* healthy and ailing individuals
* men and females
* adults and children

Exclusion Criteria:

* the participants were not be: incapacitated persons, soldiers, prisoners and persons dependent in any way from the investigators

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy people and inviduals with undiagnosed diseases or/and chronic symptoms such as: hay fever, skin and food allergies or eg. chronic fatigue.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-02-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Intestinal parasites | 1 day (single evaluation of current samples)
  The fecal samples will be assessed qualitavely in terms of life forms of parasites present in human intestine, i.e.: eggs and larvas of flukes, tapeworms and nematodes, as well as protozoa trophozoites and cysts.
Giardia antigen test | 1 day (single evalutaion of all samples through study completion)
  Stool test for Giardia lamblia antigen (ELISA kit)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sutkowy, PhD, Principal Investigator — Nicolaus Copernicus Univeristy
Locations (1):
- The Chair of Medical Biology, Collegium Medicum of Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No